CLINICAL TRIAL: NCT02831634
Title: A Feasibility Study to Identify T-cell Responses to Neo-epitopes in Tumor Invaded Lymph Nodes
Brief Title: A Feasibility Study to Identify T-cell Responses to Neo-epitopes in Tumor Invaded Lymph Nodes (NeoEpitope)
Acronym: NeoEpitope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2015-06
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Cutaneous Melanoma
Keywords: Breast cancer; cutaneous melanoma
MeSH Terms: conditions — Breast Neoplasms; Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sampling (Other)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — After inclusion in the protocol, a blood sample (50 mL in EDTA tubes) will be withdrawn during pre-operative consultation.

SUMMARY:
Feasibility study for a method allowing identification of tumor mutated epitopes in patients with breast cancer or cutaneous melanoma, and quantification of CD8+ T cells specific for these tumor neo-antigens in their lymph nodes

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years Patient with HR+ , HER2- and node-positive (proven by cytology) invasive ductal carcinoma breast cancer, grade (SBR) II or III, and having an axillary dissection programmed, Or patient having cutaneous melanoma scheduled for a lymph node dissection at the Institut Curie including dissection of the lymph nodes draining the tumor, Voluntary having signed and dated written informed consents prior to any specific study procedure,

Exclusion Criteria:

Patients treated for a breast cancer who received neoadjuvant chemotherapy Patients treated for breast cancer with distant metastases (M+)• Only for patients with breast cancer: oral or systemic corticosteroids treatment received within 30 days prior surgery Patients on immunosuppressive treatment or diagnosed of an immunodeficiency Patients with known chronic viral infection as HIV1 or 2, HBV, HCV Patients with other cancer diagnosed within 5 years (except squamous cell cutaneous carcinomas) Patients without a French social security Patients deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of a method allowing identification of tumor mutated epitopes in patients with breast cancer or cutaneous melanoma and quantification of CD8+ T cells specific for the tumor neo-antigens identified in the lymph nodes. | up to 24 months
  Feasibility study for a method allowing identification of tumor mutated epitopes : Identification of MHC cl I and II restricted tumor neo-epitopes by two different methods i.e. by an elution-HPLC method performed on cell lines derived from tumor cells obtained from invaded lymph node, or using predictive algorithms on tumor sequencing data.

SECONDARY OUTCOMES:
Quantification of CD4+ T lymphocytes specific for identified tumor neo-antigens in the lymph nodes. | up to 24 months
Quantification of CD4+ and CD8+ T lymphocytes specific for identified neo-antigens in the blood and tumor. | up to 24 months
Comparison of the frequency and relative amplitude of the T cell response specific for the tumor neo-epitopes with other immune responses and responses against known tumor antigens. | up to 24 months
  Comparison of the frequency and relative amplitude of the T cell response specific for the tumor neo-epitopes with other immune responses such as anti-viral memory responses (influenza A, ...), chronic viral responses (cytomegalovirus [CMV] Epstein-Barr virus [EBV], ...) and responses against known tumor antigens (such as NY-ESO-1, MAGE-A3, p53, gp100 ....).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).